CLINICAL TRIAL: NCT07037381
Title: A Study to Explore the Physiological Impact of AIR+ KN95 Masks on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innosparks Pte Ltd. (Industry)
Collaborators: Department of Paediatrics, Yong Loo Lin School of Medicine, National University of Singapore (Unknown); Khoo Teck Puat-National University Children's Medical Institute, National University Health System (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ISPL - PIEC/2022/050
Record Dates: First submitted 2025-06-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects
Keywords: Respiratory Protection; Physiological Impact; Particulate Respirators; KN95 Pediatric Mask; Air Pollution; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rest followed by mild exertion without mask and while wearing KN95 mask (Experimental): All study participants (single group) underwent, Rest (Reading) with no mask (control), rest (Reading) while wearing AIR+KN95 mask (intervention) followed by mild exertion without mask (control), mild exertion with the AIR+KN95 mask (intervention)
  Interventions: Other: KN95 mask

INTERVENTIONS:
Other: KN95 mask — AIR+ KN95 mask

SUMMARY:
The primary objective is to evaluate the physiological impact of AIR+ KN95 Masks on end-tidal carbon dioxide (ETCO2) of children aged 7 to 14 years of age. The secondary outcomes include other physiological parameters such as oxygen saturation (SPO2), heart rate (HR) and respiratory rate (RR). In addition, the investigators will assess the general well-being and comfort level of the child when wearing the AIR+ KN95 Mask.

DETAILED DESCRIPTION:
There is potential for severe haze episodes to occur in Singapore, and the main air pollutant in the event of haze is particulate matter (PM). Short-term exposure (continuous exposure to unhealthy daily average PSI levels over a period of a few days) to haze like the pattern seen in Singapore may cause irritation of the eyes, nose, and throat in healthy individuals. Haze particles can also affect the heart and lungs, especially in people who already have chronic heart or lung disease e.g., asthma, chronic obstructive pulmonary disease (COPD), or heart failure.

Haze is a perennial problem in Singapore. Commercially available disposable particulate respirators are typically certified for surgical and occupational use. The test standards are specified according to adult breathing conditions and fit. As commercially available disposable masks designed for occupational use are mainly for adults, such masks do not fit well on children, they do not serve well as protection against Particulate Matter 2.5 (PM 2.5), an air pollutant found in transboundary smoke haze.

Commercially available disposable particulate respirators are typically certified under the NIOSH and CE EN 149:2001+A1:2009 standards for surgical and occupational use. These respiratory masks are tested to filter particulate matter in the air with varying degrees of filtering efficiencies according to the respective categories, e.g. NIOSH KN95 certifies respirators to filter at least 95% of non-oil particulates. The test standards are specified according to adult breathing conditions and fit.

Children's respiratory minute volume and rate are different from adults. As commercially available disposable masks designed for occupational use are mainly for adults, such masks do not fit well on children, they do not serve well as protection against Particulate Matter 2.5 (PM 2.5). As haze is a perennial problem, and there is potential for severe haze episodes to occur again, there is a need to consider the development of disposable particulate respirator with enhanced safety and comfort specific for use in children.

ST Engineering Innosparks Pte. Ltd. developed a new type of disposable particulate respirator (hereon referred to as AIR+ KN95 Mask) that is suitable for use in both adults and children, from ages 7 and above. The masks come in S, M and L sizes, and have been tested according to the KN95 protocol for respirators.

Studies have shown that prolonged wearing of disposable particulate respirators may lead to an increase in carbon dioxide (CO2) levels in the dead space of the respirator as well as in the re-breathing of the expired air when wearing it. The increased CO2 levels may result in headaches, increased irritability, and breathing difficulty. In addition, there is some discomfort due to the accumulation of heat and humid air in the dead space of between the respirator and face. However, the mask design is based on our previous AIR+ Smart Mask specifications, which was previously evaluated in a clinical trial performed in collaboration with NUH and the data published in a peer-reviewed journal1, showing no significant increase in CO2 retention and the mask was found to be comfortable at rest and on mild exertion. The mask was commercially launched in 2015.

As the masks were developed specifically for school-going children, this study is designed to explore whether the new disposable particulate respirator is safe and effective for use in healthy children aged 7 to 14 years of age. This is through measuring the variation of carbon dioxide levels in children whilst wearing the AIR+ KN95 Mask. End-tidal carbon dioxide pressure (ETCO2) is a good indicator of arterial carbon dioxide pressure (PaCO2) in healthy adults and children and has been used for continuous direct assessment of PaCO2 in clinical contexts. The normal range of PaCO2 is from 35 - 45 mmHg. As there is a slight margin of difference between ETCO2 and PaCO2 values during measurement of about 1.6 +/- 4.3mmHg, this study defines 30 to 50mmHg as the acceptable range for ETCO2 levels.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 7 and 14 years of age (inclusive)
2. Subjects and their parents or legal guardian must provide their consent/ assent to take part in this study

Exclusion Criteria:

1. Subjects with any known cardiorespiratory conditions (including but not limited to the following: asthma, bronchitis, cystic fibrosis, congenital heart disease, emphysema)
2. Subjects with any known medical conditions that may be exacerbated by strenuous activity, including but not limited to the following: exercise-induced asthma, lower respiratory infection (including pneumonia, bronchitis) in the past 2 weeks, anxiety disorders, diabetes, hypertension, or epilepsy/ seizure disorder
3. Subjects with any physical disability from medical, orthopaedic, or neuromuscular disorders
4. Subjects who have an acute upper respiratory tract infection/ moderately severe rhinitis (i.e. blocked nasal passages) on the day of the study
5. Subjects who may compromise the integrity of the mask fit (e.g. those with excessive facial hair)

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
End-tidal Carbon Dioxide | Measured every minute for 24 minutes over 4 segments. 1. Rest with no mask (control)-5minutes 2. Rest with AIR+KN95 mask (intervention) -5minutes 3. Mild exertion without mask (control)-7minutes 4. Mild exertion with AIR+KN95 mask(intervention) -7minutes
  Single-use nasal cannulas used in conjunction with Nomoline™ Adapters connected to a Masimo Rad-97™ Pulse CO-Oximeter™ with NomoLine Capnography to log the End-tidal Carbon Dioxide (ETCO2), respiratory rate (RR) information, oxygen saturation (SpO2) and heart rate (HR).

SECONDARY OUTCOMES:
Oxygen Saturation | Measured every minute for 24 minutes over 4 segments. 1. Rest with no mask (control)-5minutes 2. Rest with AIR+KN95 mask (intervention) -5minutes 3. Mild exertion without mask (control)-7minutes 4. Mild exertion with AIR+KN95 mask(intervention) -7minutes
  Single-use nasal cannulas used in conjunction with Nomoline™ Adapters connected to a Masimo Rad-97™ Pulse CO-Oximeter™ with NomoLine Capnography to log the End-tidal Carbon Dioxide (ETCO2), respiratory rate (RR) information, oxygen saturation (SpO2) and heart rate (HR).
Respiratory Rate | Measured every minute for 24 minutes over 4 segments. 1. Rest with no mask (control)-5minutes 2. Rest with AIR+KN95 mask (intervention) -5minutes 3. Mild exertion without mask (control)-7minutes 4. Mild exertion with AIR+KN95 mask(intervention) -7minutes
  Single-use nasal cannulas used in conjunction with Nomoline™ Adapters connected to a Masimo Rad-97™ Pulse CO-Oximeter™ with NomoLine Capnography to log the End-tidal Carbon Dioxide (ETCO2), respiratory rate (RR) information, oxygen saturation (SpO2) and heart rate (HR).
Heart Rate | Measured every minute for 24 minutes over 4 segments. 1. Rest with no mask (control)-5minutes 2. Rest with AIR+KN95 mask (intervention) -5minutes 3. Mild exertion without mask (control)-7minutes 4. Mild exertion with AIR+KN95 mask(intervention) -7minutes
  Single-use nasal cannulas used in conjunction with Nomoline™ Adapters connected to a Masimo Rad-97™ Pulse CO-Oximeter™ with NomoLine Capnography to log the End-tidal Carbon Dioxide (ETCO2), respiratory rate (RR) information, oxygen saturation (SpO2) and heart rate (HR).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel YT Goh, MBBS, FRCPCH, Principal Investigator — Department of Paediatrics, Khoo Teck Puat - National University Children's Medical Institute, National University Hospital, Singapore
Locations (1):
- ST Engineering Innosparks Pte Ltd, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Only members of the study team e.g PI, con-investigator, and study coordinator, will have access to the data. Data collected will be de-identified and coded at source. Confidentiality of the data will be maintained at all times.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT07037381/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT07037381/ICF_001.pdf